CLINICAL TRIAL: NCT04304365
Title: Feasibility of Home Follow-up After Medication Abortion (MAB)
Brief Title: Home Follow-up After Medication Abortion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to implement the study due to delays from COVID-19 policies which postponed the start.
Sponsor: Boston Medical Center (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-39499
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Medical; Abortion, Fetus
Keywords: Home follow-up; Clinic follow-up; Low Sensitivity Pregnancy Test (LSPT); Text messaging; Medication abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic follow-up group (Active Comparator): All participants in this group will receive the standard of care at BMC which includes receiving a follow-up visit date and time before leaving the initial visit, when they receive the medications for abortion. Patients then return to clinic 1-2 weeks later to be seen by a provider with an ultrasound for confirmation of abortion completion. Participants who do not come for a return visit receive one phone call to reschedule their appointment.
  Interventions: Other: Follow-up clinic visit
- Home follow-up group (Experimental): Participants enrolled in the home follow-up group will be instructed that they will be contacted by research staff through text message 14 days after the initial visit. At enrollment, they will receive instruction for timing of contact, how to use the LSPT, as well as the test itself. The participant will take the pregnancy test at home in 14 days and answer completion questions by text message for follow-up. Patients that screen positive will be asked to return to clinic for a visit with a provider.
  Interventions: Other: Text message; Other: Low Sensitivity Pregnancy Test (LSPT)

INTERVENTIONS:
Other: Follow-up clinic visit — Participants will be scheduled for a visit with a provider in 1-2 weeks that will include an ultrasound examination.
  Arms: Clinic follow-up group
Other: Text message — Participants will be instructed that they will be contacted by research staff through text message 14 days after the initial visit. They will receive a survey link through text message at this time.
  Arms: Home follow-up group
Other: Low Sensitivity Pregnancy Test (LSPT) — Participants will be instructed on how to test their urine 14 days after the medication abortion for continued pregnancy. LSPT can detect hCG levels as low as 2000 mIU/ml.
  Arms: Home follow-up group

SUMMARY:
This study aims to evaluate a home follow-up alternative after medication abortion with pregnancy testing and a completion test. Clinical evaluation after a medication abortion (MAB) is standard of care to diagnose continued pregnancy and treat complications, typically done with a provider and an ultrasound examination or serial blood testing. Follow-up rates in the literature after MAB have been found to be 51% to 77% in recent literature using these standard follow-up methods. Though medication abortion is highly efficient, the on-going pregnancy rate is about 4% for pregnancies with gestational age up to 70 days from last menstrual period, thus highlighting the importance of follow-up as patients may not know they have a continued pregnancy weeks to even months after taking medication for an abortion. The investigators plan on providing participants with the option of a home follow-up option versus the standard of care (clinic) option. The primary objective of this study is looking at follow-up rates by each of these groups. As more options are provided for follow-up to patients, it is hoped that follow-up rates will improve and reduce the burdens of clinic visits on both providers and patients, ultimately making continued pregnancy after a medication abortion a never event.

DETAILED DESCRIPTION:
The primary objective of this research is to determine if introducing home follow-up will improve follow-up rates after medication abortion

Secondary objectives of the study are to:

* assess the feasibility of mobile phone text messaging with low sensitivity pregnancy testing for home follow-up after medication abortion
* assess the acceptability of chosen follow-up after medication abortion
* determine the complication rate, emergency room visit rate, and ongoing pregnancy rate after home follow-up

This prospective cohort study will be carried out at a single, urban hospital-based abortion clinic exploring the feasibility and acceptability of home follow-up after medication abortion with text messaging and a Low Sensitivity Pregnancy Test (LSPT). Participants will be recruited from a single abortion practice at Boston Medical Center (BMC) in Boston, Massachusetts. This clinic serves a multi-ethnic population from the South Boston area, with most patients English and Spanish speaking and covered by public insurance. Abortion care is provided by obstetrics and gynecology residents, family planning fellows, nurse practitioners, and family planning doctors.

As part of the study participants will be given the choice to have clinic follow-up or home follow-up. The clinic follow-up cohort will receive our clinic standard of care - they will be scheduled for a visit with a provider in 1-2 weeks that will include an ultrasound examination. This cohort will be asked the same questions to assess completion that will be asked of the home follow-up group.

Participants enrolled in the home follow-up group will be instructed that they will be contacted by research staff through text message 14 days after the initial visit. At enrollment, they will receive instruction for when the study team will be contacting them, how to use the LSPT, as well as the test itself. The participant will take the pregnancy test at home in 14 days and answer completion questions by text message for follow-up. Patients that screen positive will be asked to return to clinic for a visit with a provider.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speakers
* Have a working phone they consider their own with text messaging capabilities
* Have a viable intrauterine pregnancy
* Are eligible for a medication abortion (10 weeks gestational age or less)
* Elect the method of medication abortion

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Completed follow-up for the clinic group | 2 weeks
  Percent of participants in this group that return to the scheduled clinic visit
Completed follow-up for the home group | 2 weeks
  Percent of participants in this group that completed the final texted survey

SECONDARY OUTCOMES:
Any follow up | 42 days
  Number of participants who had any follow-up based on unscheduled clinic visits
Ongoing pregnancy | 42 days
  Number of participants found to have an ongoing pregnancy after a medication abortion
Complications after the medical abortion | 42 days
  Number of participants presenting with complications such need for transfusion and treatment of a uterine infection
Number of emergency visits | 42 days
  Number of participants presenting to the emergency room
Acceptability of chosen follow-up | 2 weeks
  An investigator developed survey will document acceptability of the follow-up process, given at the follow-up visit
Screen positive for pregnancy in the home follow-up group | 2 weeks
  The percentage of participants that screen positive from a urine test using LSPT in the home follow-up group, requiring a clinic follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Cara Delaney, MD, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No